CLINICAL TRIAL: NCT00805285
Title: Oral Budesonide and Rectal Hydrocortisone for the Treatment of Extensive Ulcerative Colitis: A Pilot Study
Brief Title: The Use of Oral Budesonide and Rectal Hydrocortisone for the Treatment of Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to insufficient enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Raymond Cross, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30365
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Ulcerative Colitis; Budesonide; Corticosteroids
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Oral Budesonide and Rectal Hydrocortisone (Experimental): See intervention
  Interventions: Drug: Combination Oral Budesonide and Rectal Hydrocortisone

INTERVENTIONS:
Drug: Combination Oral Budesonide and Rectal Hydrocortisone — Budesonide 9 mg PO (oral) daily and hydrocortisone 100 mL PR (enema) for an 8-week period. The doses of each drug to be used in the pilot study are standard doses used in clinical practice. After 8-weeks, the budesonide will be tapered in the following manner: 1) budesonide 6 mg PO daily and hydrocortisone 100 ml PR every other day (EOD) for 3 weeks then 2) budesonide 3 mg PO daily and hydrocortisone 100 ml PR 2 x per week for 3 weeks then 3) discontinue budesonide.
  Other Names: Entocort

SUMMARY:
The purpose of this study is to evaluate if the combination of oral budesonide and rectal hydrocortisone improves symptoms in patients with active ulcerative colitis. Also, we would like to determine if oral budesonide and rectal hydrocortisone has fewer and less severe side effects compared to standard steroids (prednisone).

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a common chronic inflammatory condition of the intestines that results in bloody diarrhea, abdominal pain, and extraintestinal manifestations of disease. The disease course is typically chronic, characterized by periodic exacerbations followed by symptom- free intervals; less commonly symptoms are continuous and unrelenting. The symptoms and disease course have a profound, detrimental impact on the quality of life in patients with UC.

The initial therapeutic approach depends upon both the extent of colonic involvement and the severity of the disease process at presentation. Typically, patients are treated based on a pyramid or "Step up" approach. If patients have mild symptoms, they receive less powerful therapies lower in the pyramid with fewer side effects. Patients with disease confined to distal colon are typically treated with topical therapies including either 5-ASA or steroid enemas. However, as symptoms worsen or if severe at the time of diagnosis, patients receive more aggressive therapies higher in the pyramid including steroids. Despite medical therapy, 50% will have colectomy or become steroid dependent one year after receiving steroids.

Steroids are associated with significant side effects. Adverse consequences of steroids are related to dose and duration of exposure, and include but are not limited to cosmetic side effects, ocular disease (glaucoma, cataracts), diabetes, hypertension, vascular disease, osteoporosis, neuropsychiatric complications, and increased risk of infection.

Newer "designer" corticosteroids including budesonide have reduced systemic bioavailability and high local anti-inflammatory activity; as a result it is associated with fewer and less severe side effects. Studies have proven the efficacy of budesonide in inducing remission in active Crohn's disease. However, the data for the use of oral budesonide in patients with UC is less extensive. However, the data regarding the efficacy of topical therapy for left-sided UC is extensive. Randomized controlled trials of budesonide enemas have demonstrated similar efficacy and safety profile to hydrocortisone enemas in the induction of remission of left sided UC. We have chosen to utilize hydrocortisone enemas in our study as it is widely available in the United States.

A 52-week open-label pilot study will be performed at the University of Maryland Medical Center. Subjects will include patients with previously or newly diagnosed extensive ulcerative colitis. Patients will be treated with oral budesonide and rectal hydrocortisone for 8 weeks followed by a predetermined taper. All patients will undergo research clinic visits at enrollment and week 8. During these visits, patients will complete a series of questionnaires that measure the patient's disease activity, quality of life, side effects, medical compliance, and other parameters. Blood draws and stool studies are required at each study visit to monitor blood counts, electrolytes, liver function, inflammatory markers, and adrenal function. Additionally, at week 16, an ACTH (cosyntropin) stimulation test will be performed. After obtaining a basal cortisol level, 250 ug of cosyntropin is given intravenously. Plasma samples of cortisol will then be drawn at 30 minutes to assess for adrenal insufficiency. Close follow-up with eight 30-min telephone sessions (every 2-3 weeks) will also be conducted to assess disease activity and adverse events.

The goal of this study is to determine whether combination therapy using oral budesonide and topical hydrocortisone will result in the induction of remission in patients with active extensive ulcerative colitis. Further, we aim to show that combination therapy is better tolerated and has less severe side effects compared to conventional therapy with prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Written, voluntary, informed consent given
* 18 years or older
* Speak and read English
* Extensive ulcerative colitis based upon endoscopy, histopathology, and clinical symptoms
* SCCAI Score > 3
* Presence of diarrhea (3 or more bowel movements per 24 hours) AND grossly visible blood in stool

Exclusion Criteria:

* Serum creatinine > 2.0 mg/dL
* Pregnant or breastfeeding
* Prior history of total or subtotal colectomy, or currently has an ostomy
* History or suspicion of Crohn's disease or Indeterminate colitis
* Diagnosis of any condition deemed by the investigator inhibiting completion of the trial
* Initiated therapy with or change in mesalamine dose within the last 4 weeks
* Change in azathioprine, 6-mercaptopurine, or cyclosporine within the last 8 weeks
* Currently taking or have used corticosteroids within the last 8 weeks
* Rectally administered mesalamine or steroids within the last 2 weeks
* Current or prior use of anti-TNF alpha agents within the last 8 weeks
* Experimental ulcerative colitis agents within the last 8 weeks
* Concomitant use of CYP3A4 activity inhibitor (e.g. ketoconazole, itraconazole, ritonavir, indinavir, erythromycin)
* Uncontrolled diabetes (HgA1c > 8.0) within 1 year
* Unstable Coronary artery disease/Class III/IV CHF
* Decompensated cirrhosis (e.g. encephalopathy, renal failure, ascites, GIB)
* Any known infection requiring antibiotics
* Active Clostridium difficile infection
* COPD requiring home oxygen
* HIV/AIDS with CD4 < 200 or AIDs-defining illnesses/infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond K Cross, MD, MS, Principal Investigator — University of Maryland, College Park; Leyla J Ghazi, MD, Study Chair — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Oral Budesonide and Rectal Hydrocortisone: Budesonide 9 mg po daily and Rectal Hydrocortisone once daily
Period: Overall Study
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: The only enrolled patient was withdrawn secondary to disease worsening.
Groups:
- Combination Oral Budesonide and Rectal Hydrocortisone: Intervention Arm
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Simple Clinical Colitis Disease Activity (SCCAI)
Description: Scores range from 0-19. Higher scores indicated increased disease severity. A score less than 3 is consistent with clinical remission.
Time Frame: 0, 2, 4, 6, and 8 weeks
Population: The only patient enrolled withdrew; there was no data to analyze.
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 0

2. Primary Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Description: Scores range from 10-70 where higher scores indicated better quality of life.
Time Frame: Week 0 and 8
Population: The only patient enrolled withdrew; there was no data to analyze.
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 0

3. Secondary Outcome: ACTH Stimulation Test
Description: An increase in cortisol after stimulation by ACTH is normal. Blood cortisol after ACTH stimulation should be greater than 18 - 20 mcg/dL, depending on the dose of cosyntropin used.
Time Frame: Week 16
Population: The only patient enrolled withdrew; there was no data to analyze.
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 0

4. Secondary Outcome: Adverse Events
Time Frame: 0, 2, 4, 6, 8, 11, 14, 20, 26, and 52 weeks
Measure: Number; unit: Adverse events
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 1
Adverse events | 2

5. Secondary Outcome: C Reactive Protein
Description: Higher values indicated increased disease activity
Time Frame: Week 0 and 8
Population: The only patient enrolled withdrew; there was no data to analyze.
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Combination Oral Budesonide and Rectal Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Oral Budesonide and Rectal Hydrocortisone (N=1)
Worsening of ulcerative colitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Oral Budesonide and Rectal Hydrocortisone (N=1)
Portal vein and superior mesenteric vein thrombosis (Vascular disorders) | 1 — The only enrolled patient was found to have a portal and superior mesenteric vein thrombosis. This was thought to be related to the underlying ulcerative colitis and not related to the intervention.

LIMITATIONS AND CAVEATS:
The study was terminated early by the University of Maryland HRPO secondary to limited recruitment of participants. This resulted in an inability to analyze the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No